CLINICAL TRIAL: NCT03394365
Title: Multicenter, Open-Label, Phase 3 Study of Tabelecleucel for Solid Organ or Allogeneic Hematopoietic Cell Transplant Subjects With Epstein-Barr Virus-Associated Post-Transplant Lymphoproliferative Disease After Failure of Rituximab or Rituximab and Chemotherapy
Brief Title: A Phase 3 Study of Tabelecleucel for Participants With Epstein-Barr Virus-Associated Post-Transplant Lymphoproliferative Disease After Failure With Rituximab or Rituximab and Chemotherapy
Acronym: ALLELE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATA129-EBV-302/F60085DL302; 2024-516622-57-00 (EU CTIS Number); NCT03392142 (obsolete NCT alias)
Record Dates: First submitted 2017-12-29; First posted 2018-01-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Epstein-Barr Virus+ Associated Post-transplant Lymphoproliferative Disease (EBV+ PTLD); Solid Organ Transplant Complications; Lymphoproliferative Disorders; Allogeneic Hematopoietic Cell Transplant; Stem Cell Transplant Complications
Keywords: Epstein-Barr Virus (EBV)-associated Lymphoproliferative Disease (LPD); Epstein-Barr Virus (EBV); Cytotoxic T lymphocyte (CTL); Cancer After Transplant; Kidney transplant; Renal transplant; Liver transplant; Heart transplant; Lung transplant; Intestinal transplant; Pancreas transplant; Post-transplant Lymphoma; Solid Organ Transplant (SOT); Bone Marrow Transplant Complications; Epstein-Barr Virus-specific Cytotoxic T Lymphocytes (EBV-CTL); Hematopoietic Cell Transplant (HCT); Hematopoietic Stem Cell Transplantation (HSCT); Allogeneic Hematopoietic Cell Transplant; Allogeneic, Off-The-Shelf T-cell Immunotherapy
MeSH Terms: conditions — Lymphoproliferative Disorders; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort SOT-R (C-SOT-R) (Experimental): Participants with EBV+ PTLD following SOT that has failed rituximab will receive IV tabelecleucel.
  Interventions: Biological: tabelecleucel
- Cohort SOT-R+C (C-SOT-R+C) (Experimental): Participants with EBV+ PTLD following SOT that has failed both rituximab and chemotherapy will receive IV tabelecleucel.
  Interventions: Biological: tabelecleucel
- Cohort HCT (C-HCT) (Experimental): Participants with EBV+ PTLD following HCT that has failed rituximab containing regimen will receive IV tabelecleucel.
  Interventions: Biological: tabelecleucel

INTERVENTIONS:
Biological: tabelecleucel — Tabelecleucel is being investigated as an off-the-shelf, allogeneic T-cell immunotherapy for the treatment of EBV+ malignancies and diseases.
  Other Names: tab-cel®; ATA129; EBV-CTL; Ebvallo®

SUMMARY:
The purpose of this study is to determine the clinical benefit and characterize the safety profile of tabelecleucel for the treatment of Epstein-Barr virus-associated post-transplant lymphoproliferative disease (EBV+ PTLD) in the setting of (1) solid organ transplant (SOT) after failure of rituximab (SOT-R) and rituximab plus chemotherapy (SOT-R+C) or (2) allogeneic hematopoietic cell transplant (HCT) after failure of rituximab.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase 3 study to assess the efficacy and safety of tabelecleucel for the treatment of EBV+ PTLD in the setting of SOT-R and SOT-R+C (Cohort [C]-SOT) or HCT after failure of rituximab (C-HCT).

SOT-R further included participants:

1. who did not receive chemotherapy and did not have a documented medical reason not to receive chemotherapy (SOT-Ro) or
2. who were considered chemotherapy ineligible/inappropriate (SOT-R-Ci)

Combined population (SOT-R-Ci, SOT-R+C, and HCT) and (SOT-R-Ci and SOT-R+C) who received commercial product, or a product manufactured using a comparable process version (PV) were also used for analysis of outcomes.

Enrollment will be preceded by confirmation of availability of partially human leukocyte antigen (HLA) matched and restricted tabelecleucel for the participant.

Study procedures and product administration will be the same for each cohort. Tabelecleucel will be administered in cycles lasting 5 weeks (35 days). During each cycle, participants will receive intravenous tabelecleucel at a dose of 2 × 10^6 cells/kg on Days 1, 8, and 15, followed by observation through Day 35. Treatment will continue until maximal response, unacceptable toxicity, initiation of non protocol therapy, or failure of tabelecleucel with up to 2 different HLA restrictions (C-SOT) or up to 4 different HLA restrictions (C-HCT). The study includes a total of 5 years of follow-up for disease and survival status for participants enrolled before or after 09 October 2023 to reach the initial sample size of 33 participants in both cohorts. For all other participants enrolled after 09 October 2023 and after the initial sample of 33 participants in both cohorts has been reached in both cohorts, the follow-up will be every 3 months, up to 12 months, as assessed on anniversary of Cycle 1 Day 1. For responders, the follow-up will be 12 months from the date of initial response.

ELIGIBILITY:
Inclusion Criteria:

1. Prior SOT of kidney, liver, heart, lung, pancreas, small bowel, or any combination of these (C-SOT); or prior allogeneic HCT (C-HCT).
2. A diagnosis of locally assessed, biopsy-proven EBV+ PTLD.
3. Availability of appropriate partially HLA-matched and restricted tabelecleucel has been confirmed by the sponsor.
4. Measurable, 18F-deoxyglucose (FDG)-avid (Deauville score ≥ 3) systemic disease using Lugano Classification response criteria by positron emission tomography (PET)-diagnostic computed tomography (CT), except when contraindicated or mandated by local practice, then magnetic resonance imaging (MRI) may be used. For participants with treated central nervous system (CNS) disease, a head CT and/or brain/spinal MRI as clinically appropriate will be required to follow CNS disease response per Lugano Classification response criteria.
5. Treatment failure of rituximab or interchangeable commercially available biosimilar monotherapy (C-SOT-R or C-HCT) or rituximab plus any concurrent or sequentially administered chemotherapy regimen (C-SOT-R+C) for treatment of PTLD.
6. Males and females of any age.
7. Eastern Cooperative Oncology Group performance status ≤ 3 for participants aged ≥ 16 years; Lansky score ≥ 20 for participants < 16 years.
8. For C-HCT only: If allogeneic HCT was performed as treatment for an acute lymphoid or myeloid malignancy, the underlying primary disease for which the participant underwent transplant must be in morphologic remission.
9. Adequate organ function.

   1. Absolute neutrophil count ≥ 1000/μL, (C-SOT) or ≥ 500/μL (C-HCT), with or without cytokine support.
   2. Platelet count ≥ 50,000/μL, with or without transfusion or cytokine support. For C-HCT, platelet count < 50,000/μL but ≥ 20,000/μL, with or without transfusion support, is permissible if the participant has not had grade ≥ 2 bleeding in the prior 4 weeks (where grading of the bleeding is determined per the National Cancer Institute's Common Terminology Criteria for Adverse Events [CTCAE], version 5.0).
   3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin each < 5 × the upper limit of normal; however, ALT, AST, and total bilirubin each ≤ 10 × upper limit of normal is acceptable if the elevation is considered by the investigator to be due to EBV and/or PTLD involvement of the liver as long as there is no known evidence of significant liver dysfunction.
10. Participant or participant's representative is willing and able to provide written informed consent.

Exclusion Criteria:

1. Currently active Burkitt, T-cell, NK/T-cell lymphoma/LPD, Hodgkin, plasmablastic, transformed lymphoma, active hemophagocytic lymphohistiocytosis, or other malignancies requiring systemic therapy.
2. Daily steroids of > 0.5 mg/kg prednisone or glucocorticoid equivalent, ongoing methotrexate, or extracorporeal photopheresis.
3. Untreated CNS PTLD or CNS PTLD for which the participant is actively receiving CNS-directed chemotherapy (systemic or intrathecal) or radiotherapy at enrollment. NOTE: Participants with previously treated CNS PTLD may enroll if CNS-directed therapy is complete.
4. Suspected or confirmed grade ≥ 2 graft-versus-host disease (GvHD) per the Center for International Blood and Marrow Transplant Research consensus grading system at enrollment.
5. Ongoing or recent use of a checkpoint inhibitor agent (eg, ipilimumab, pembrolizumab, nivolumab) within 3 drug half-lives from the most recent dose to enrollment.
6. For C-HCT: active adenovirus viremia.
7. Need for vasopressor or ventilatory support.
8. Antithymocyte globulin or similar anti-T cell antibody therapy ≤ 4 weeks prior to enrollment.
9. Treatment with Epstein-Barr virus cytotoxic T lymphocytes or chimeric antigen receptor T cells directed against B cells within 8 weeks of enrollment (C-SOT or C-HCT), or unselected donor lymphocyte infusion within 8 weeks of enrollment (C-HCT only).
10. Female who is breastfeeding or pregnant or female of childbearing potential or male with a female partner of childbearing potential unwilling to use a highly effective method of contraception.
11. Inability to comply with study-related procedures.
12. Any medical condition or organ system dysfunction that in the investigator';s opinion, could compromise the participant's safety or ability to complete the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2017-12-29 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) in the Analysis Cohorts C-SOT, C-HCT, and Combined Population (C-SOT-R+C, C-SOT-R-Ci, and C-HCT) Who Received Commercial Product, or a Product Manufactured Using a Comparable PV | 2 years

SECONDARY OUTCOMES:
Duration of Response (DOR) in the Analysis Cohorts C-SOT and C-HCT Separately | 2 years
ORR in the Analysis Cohorts C-SOT and C-HCT Combined | 2 years
ORR and DOR in Participants who Received Commercial Product or a Product Manufactured Using a Comparable PV in the Analysis Cohorts C-SOT-R-Ci and C-SOT-R+C Separately and Combined, and in the Analysis Cohort C-HCT | 2 years
DOR in a Combined Population (SOT-R-Ci, SOT-R+C, and HCT) who Received Commercial Product or a Product Manufactured Using a Comparable PV | 2 years
Rates of Complete Response (CR) and Partial Response (PR) | 2 years
Time to Response | 2 years
Time to Best Response | 2 years
Overall Survival (OS) | 2 years
Rates of Allograft Loss or Rejection Episodes (Analysis Cohort C-SOT) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Anke Friedetzky, Study Director — Pierre Fabre Laboratories
Locations (71):
- United States (40):
  - City of Hope (Adults and Pediatrics), Duarte, California
  - University of California San Diego Moores Cancer Center (Adults only), La Jolla, California
  - Loma Linda University Medical Center (Adults only), Loma Linda, California
  - Children's Hospital Los Angeles, Div. of Research Immunology/BMT (Adults and Pediatrics), Los Angeles, California
  - UCLA Medical Center (Adults and Pediatrics), Los Angeles, California
  - University of California Davis Comprehensive Cancer Center (Adults only), Sacramento, California
  - Yale University (Adults and Pediatrics), New Haven, Connecticut
  - MedStar Georgetown University Hospital (Adults and Pediatrics), Washington D.C., District of Columbia
  - University of Florida (Adults and Pediatrics), Gainesville, Florida
  - University of Miami/Jackson Memorial Hospital (Adults only), Miami, Florida
  - Winship Cancer Institute (Adults only), Atlanta, Georgia
  - Arthur M. Blank Hospital (Pediatrics), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago (Adults and Pediatrics), Chicago, Illinois
  - University of Chicago Medical Center - Duchossois Center for Advanced Medicine (Adults only), Chicago, Illinois
  - Loyola University Medical Center (Adults and Pediatrics), Maywood, Illinois
  - University of Maryland School of Medicine (Adults only), Baltimore, Maryland
  - Dana Farber Cancer Institute, Brigham and Women's Hospital (Adults and Pediatrics), Boston, Massachusetts
  - Washington University School of Medicine (Adults only), St Louis, Missouri
  - Weill Cornell Medicine (Adults only), New York, New York
  - Columbia University Medical Center (Adults and Pediatrics), New York, New York
  - Memorial Sloan Kettering Cancer Center (Adults and Pediatrics), New York, New York
  - Montefiore Medical Center (Adults only), The Bronx, New York
  - Montefiore Medical Center (Pediatrics only), The Bronx, New York
  - University of North Carolina at Chapel Hill, Lineberger Comprehensive Cancer Center (Adults and Pediatrics), Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Children's Hospital (Adults and Pediatrics), Charlotte, North Carolina
  - Duke Cancer Institute (Adults and Pediatrics), Durham, North Carolina
  - Cleveland Clinic Foundation (Adults and Pediatrics), Cleveland, Ohio
  - Nationwide Children's Hospital (Pediatrics only), Columbus, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute (Adults and Pediatrics), Columbus, Ohio
  - Oregon Health and Science University Physicians Pavilion (Adults and Pediatrics), Portland, Oregon
  - Hospital of the University of Pennsylvania (Adults only), Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia Oncology Division, Blood & Marrow Transplant Section (Pediatrics), Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (Adults only), Pittsburgh, Pennsylvania
  - Medical University of South Carolina (Adults and Pediatrics), Charleston, South Carolina
  - Saint Jude Children's Research Hospital (Pediatrics only), Memphis, Tennessee
  - Vanderbilt University Medical Center Henry-Joyce Cancer Clinic (Adults and Pediatrics), Nashville, Tennessee
  - Baylor Scott and White Research Institute (Adults only), Dallas, Texas
  - University of Texas Southwestern Medical Center - Children's Medical Center (Pediatrics only), Dallas, Texas
  - MD Anderson Cancer Center (Pediatrics and Adult), Houston, Texas
  - Froedtert and Medical College of Wisconsin - Clinical Cancer Center (Adults only), Milwaukee, Wisconsin
- Australia (6):
  - The Children's Hospital at Westmead (Pediatrics only), Westmead, New South Wales
  - Westmead Hospital (Adults only), Westmead, New South Wales
  - The Prince Charles Hospital (Adults only), Chermside, Queensland
  - Royal Adelaide Hospital (Adults only), Adelaide, South Australia
  - The Royal Children's Hospital Melbourne (Pediatrics only), Melbourne, Victoria
  - Fiona Stanley Hospital (Adults only), Murdoch, Western Australia
- Medizinische Universitat Wien (Adults only), Vienna, Austria, Austria
- Belgium (2):
  - Centre Hospitalier Universitaire de Liège Site Sart Tilman (Adults and Pediatrics), Liège, Brussels Capital
  - Universitair Ziekenhuis Leuven (Adults and Pediatrics), Leuven, Flemish Brabant
- Canada (3):
  - Alberta Children's Hospital (Adults and Pediatrics), Calgary, Alberta
  - Sick Kids (Pediatrics only), Toronto, Ontario
  - Princess Margaret Cancer Centre (Adults only), Toronto, Ontario
- France (5):
  - Centre Hospitalier Universitaire de Bordeaux (Adults only), Pessac, Aquitaine
  - Centre Hospitalier Régional Universitaire de Lille (Adults and Pediatrics), Lille, Hauts-de-France
  - Hôpital Necker-Enfants Malades (Pediatrics only), Paris, Île-de-France Region
  - Hôpital Saint Antoine (Adults only), Paris, Île-de-France Region
  - Hôpital Universitaire Pitié Salpêtrière (Adults only), Paris, Île-de-France Region
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda (Adults only), Milan, Milano
  - Fondazione IRCCS Policlinico San Matteo (Adults and Pediatrics), Pavia, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli (Adults only), Roma, Roma
  - Ospedale Pediatrico Bambino Gesu (Pediatrics only), Roma, Roma
  - Azienda Ospedaliera - Universitaria Città della Salute e della Scienza di Torino (Adults only), Torino, Torino
- Spain (6):
  - Hospital Duran i Reynals (Adults and Pediatrics), Badalona, BARCELONA
  - Hospital Universitari Vall d'Hebrón - Institut de Recerca (Adults and Pediatrics), Barcelona, Barcelona
  - Hospital Universitario Marqués de Valdecilla (Adults and Pediatrics), Santander, Cantabria
  - Hospital General Universitario Gregorio Marañón (Adults and Pediatrics), Madrid, Madrid
  - University Hospital Virgen del Rocio (Adults and Pediatrics), Seville, Spain
  - Hospital Universitario La Fe (Adults and Pediatrics), Valencia, Valencia
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust (Adults only), Birmingham, England
  - King's College Hospital NHS Foundation Trust (Adults only), London, England
  - Imperial College Healthcare NHS Trust (Adults only), London, England

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahadeo KM, Baiocchi R, Beitinjaneh A, Chaganti S, Choquet S, Dierickx D, Dinavahi R, Duan X, Gamelin L, Ghobadi A, Guzman-Becerra N, Joshi M, Mehta A, Navarro WH, Nikiforow S, O'Reilly RJ, Reshef R, Ruiz F, Spindler T, Prockop S. Tabelecleucel for allogeneic haematopoietic stem-cell or solid organ transplant recipients with Epstein-Barr virus-positive post-transplant lymphoproliferative disease after failure of rituximab or rituximab and chemotherapy (ALLELE): a phase 3, multicentre, open-label trial. Lancet Oncol. 2024 Mar;25(3):376-387. doi: 10.1016/S1470-2045(23)00649-6. Epub 2024 Jan 31. PMID 38309282